CLINICAL TRIAL: NCT06464770
Title: Optimizing Infection Prophylaxis Prior to Shoulder Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jason Hsu, Associate Professor, Orthopaedic Surgery and Sports Medicine, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00020250
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Arthroplasty Shoulder; Periprosthetic Joint Infection
Keywords: periprosthetic joint infection; cutibacterium; shoulder arthroplasty; chlorhexidine
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Intervention Model Description: Randomization Option 1: Right shoulder, Test Group ; Left shoulder, Control Group Randomization Option 2: Right shoulder, Control Group ; Left shoulder, Test Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Randomization Option 1 (Experimental): Right shoulder, Test Group ; Left shoulder, Control Group
  Interventions: Drug: Chlorhexidine Gluconate
- Randomization Option 2 (Experimental): Right shoulder, Control Group ; Left shoulder, Test Group
  Interventions: Drug: Chlorhexidine Gluconate

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — Test Group: the participant's shoulder skin will be treated by the study team with the standard chlorhexidine wash at lower pressure (similar to a gentle wipe) for 30 seconds Control Group: the participant's shoulder skin will be treated by the study team with the standard chlorhexidine wash at higher pressure (similar to a massage) for 30 seconds

SUMMARY:
The goal of this interventional study is to determine the amount of skin C. acnes reduction with increased pressure during the chlorhexidine gluconate, brand name ChloraPrep, application. The main question it aims to answer is:

Does changing the pressure applied during the ChloraPrep application impact the amount of C. acnes bacteria on the skin after one hour? Researchers will compare ChloraPrep applied at a pressure similar to a gentle wipe to ChloraPrep applied at a pressure similar to a massage to see if wash the amount of C. acnes on the skin after one hour is different.

Participants will have one shoulder washed with ChloraPrep using pressure meant to impact the dermal layer, similar to a gentle wipe, and the other shoulder washed with ChloraPrep using pressure meant to impact the subdermal layer, similar to a massage. Participants will have swabs taken of their skin before the ChloraPrep application and again one hour after application to look for the amount of C. acnes on the skin.

ELIGIBILITY:
Inclusion Criteria:

* English speaking

Exclusion Criteria:

* Self report very sensitive skin
* Allergic to chlorhexidine
* Used antibiotics in the last three months
* Used acne treatment in the last three months
* Wounds on your shoulders

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Quadrants on Culture Plate of Cutibacterium Growth After ChloraPrep Application with Dermal Pressure | 60 Minutes After ChloraPrep Wash
Number of Quadrants on Culture Plate of Cutibacterium Growth After ChloraPrep Application with Subdermal Pressure | 60 Minutes After ChloraPrep Wash

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hsu, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No